CLINICAL TRIAL: NCT01335880
Title: Helping People to Exercise Regularly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS10-385
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2011-07

CONDITIONS: Obesity; Heart Disease
Keywords: Obesity; Heart Disease; Seniors; Elderly; Chronic Disease; Prevention
MeSH Terms: conditions — Obesity; Heart Diseases; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promotion I (Active Comparator): Three month time horizon
  Interventions: Behavioral: Coupons for use within the next 3 months
- Promotion II (Experimental): One week time horizon
  Interventions: Behavioral: Coupons for use within the next week

INTERVENTIONS:
Behavioral: Coupons for use within the next week — Participants who attend an exercise class will receive a coupon for a free exercise class to be used within the next week.
  Arms: Promotion II
Behavioral: Coupons for use within the next 3 months — Participants who attend an exercise class will receive a coupon to attend an exercise class for free within the next 3 months.
  Arms: Promotion I

SUMMARY:
This study tests two different incentive mechanisms to induce members of a particular urban senior center to attend more exercise classes. Coupons for future use are given to participants who attend an exercise class and will be redeemable within either a one week or three month time period, depending on which experimental group the participant is assigned to. Frequency of exercise class attendance at the end of 2 months will be the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* Member of the Philadelphia Senior Center

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Frequency of exercise class attendance | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Erte Xiao, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States